CLINICAL TRIAL: NCT05359107
Title: A Pragmatic Randomised Control Trial Comparing the Efficacy of the "Free From Pain Exercise Book" Versus "The Back Book" in Decreasing Back Pain in Adults Over 60 Years of Age.
Brief Title: The "Free From Pain Exercise Book" Versus "The Back Book".
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Talita Cumi Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FFPETFETS006
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Sarcopenia; Back Pain; Arthritis
MeSH Terms: conditions — Sarcopenia; Back Pain; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "The Free From Pain Exercise Book" (Experimental): Participants who consent and are randomised into Group 1 (experimental group) will be provided with the "Free From Pain Exercise Book". Participants in Group 1 will be asked to independently engage in the exercises included in the book throughout the entire 6 month study period. They will be advised to either do all 3 sets of exercises 3 times a week or to do the neck and low back exercises twice a week and the Otago exercises 3 times a week. The exercises should take around an hour to complete each day.
  Furthermore, it will be recommended that participants in this group read one information chapter and one metaphor each week for 12 weeks, to ensure that they absorb the information fully and do not overbear themselves with information.
  Interventions: Behavioral: "The Free From Pain Exercise Book"
- "The Back Book" (Active Comparator): Participants who consent and are randomised into Group 2 (control group) will be provided with "The Back Book". Participants in Group 2 will be asked to ensure that they read the book in its entirety during the 12-week intervention period and refer to relevant sections during the follow-up period for advice if required.
  Interventions: Behavioral: "The Back Book"

INTERVENTIONS:
Behavioral: "The Free From Pain Exercise Book" — Contains educational information and exercises to improve musculoskeletal pain and reduce sarcopenia.
  Arms: "The Free From Pain Exercise Book"
Behavioral: "The Back Book" — Contains advice and guidance on how to deal with and reduce back pain.
  Arms: "The Back Book"

SUMMARY:
This pragmatic randomised control feasibility trial aims to investigate the effectiveness of the "Free From Pain Exercise Book" in comparison to "The Back Book" for reducing back pain in adults aged 60 and over. The "Free From Pain Exercise Book" contains a 12-week exercise and education programme. The programme is designed to reduce early osteoarthritic and generalised musculoskeletal pain and fear of falling in people over the age of 60. The study will compare the effects of the Free from Pain programme when engaged in independently versus the provision of "The Back Book", which is a booklet that promotes physical activity and a reduction of sedentary behaviour for the purpose of reducing back pain.

DETAILED DESCRIPTION:
Chronic musculoskeletal conditions are the leading cause of disability worldwide. The World Health Organization estimates that approximately 1.71 billion people have musculoskeletal conditions globally. They cause a significant economic burden on the NHS, with £5 billion of England's yearly NHS budget going towards the treatment of musculoskeletal conditions. The most reported musculoskeletal ailment throughout the world is back pain, for which the lifetime prevalence has been reported to be as high as 84%. Back pain can affect individuals of all ages, but has a particularly negative effect on elderly people, causing difficulty in daily living tasks for those over 65 years old. Difficulty in completing everyday tasks can result in immobility, causing a loss of muscle mass and fitness, an increased risk of falls, further injury, and diseases associated with inactivity or sedentary behaviours (such as heart attack and some cancers).

"The Back Book" is a booklet that promotes physical activity and a reduction of sedentary behaviour for the purpose of reducing back pain. One study by Hass et, al. found that the addition of this book to standard treatment improved disability scores significantly. The use of "The Back Book" was further supported by a cluster, randomised control trial which focussed on elderly adults from nursing homes. The study found a significant improvement in disability after one month of being provided with the book. It is known that, in later life, exercise can have many physiological and psychological benefits and can improve functional ability and well-being whilst reducing illness.

The complete "Free From Pain Exercise Book" presents exercises and educational information to improve pain, strength and quality of life in seniors. The "Free from Pain" exercise programme described within the exercise book is a 12-week exercise programme. It is fusion of three different generally accepted exercise programmes. Therapeutic exercise programmes exist for individual body parts, but there is no single generalised exercise programme that targets all body parts. Hence, the creation of this fusion of programmes. The three programmes are the Otago exercises for lower body strength and balance, the motor control exercises for the lower back and the isometric exercises for the neck and shoulder.

The Otago exercise program (OEP) was developed by Robertson and Campbell for the New Zealand accident compensation corporation (ACC). The initial aim of the programme was to improve balance and strength in patients to prevent falls. Further research has shown that the Otago exercise programme is an effective intervention for coping with musculoskeletal pain in community-dwelling older adults. For treating and preventing low back pain, exercise regimes include stretching, strengthening, endurance, aerobic fitness, walking, yoga, Pilates, and motor control exercises. Among these different modalities of exercises for the rehabilitation of low back pain, motor control exercises are one of the most commonly used interventions that have proven to be beneficial. With regards to neck pain, exercise regimes vary from stretching to strengthening exercises. Among the varied regimes, isometric and strengthening exercises of the neck and shoulder are effective modalities for treating neck pain.

Alongside descriptions and images of the exercises described previously, the exercise book also contains 13 chapters. The first chapter acts as an introduction and each of the remaining 12 chapters provide a 'reason to exercise' and an 'exercise-related metaphor'. Each chapter is assigned to a week, from week 1 through to week 12. The reader is encouraged to read one chapter each week over the 12 weeks in the order that they appear in the book.

This pragmatic randomised control feasibility trial will be conducted over 6 months.

60 participants will be split into two even groups of 30 (Group 1 and Group 2). Group 1 (experimental group) will test the use of the "Free From Pain Exercise Book" for reducing back pain and improving quality of life, whilst Group 2 (control group) will test the use of "The Back Book". Each participant will be in the study for a period of six months. As the "Free From Pain" programme is a 12-week exercise programme, the first 12 weeks of the entire six-month study is defined as the intervention period. The subsequent follow-up period, which will run from the 12-week point until the six-month point, is included in the study to allow analysis of long-term participant compliance and to assess the extended effects of both the "Free From Pain Exercise Book" and "The Back Book". Participants will be asked to provide data in the form of completed surveys three times; at baseline, at 12 weeks (once the intervention period is complete) and at six months (at the end of the follow-up period). The study aims to investigate the effectiveness of the "Free From Pain Exercise Book" in comparison to "The Back Book" for reducing back pain in adults aged 60 and over. It will compare the effects of the Free from Pain programme when engaged in independently versus the provision of "The Back Book" - a booklet that promotes physical activity and a reduction of sedentary behaviour for the purpose of reducing back pain.

ELIGIBILITY:
Inclusion Criteria:

* > 60 years of age
* Has back pain

Exclusion Criteria:

* Lacking the physical ability or cardiovascular fitness required to participate in the "Free From Pain" exercises. This criterion will be explained on the participant information sheet by stating, "If you are unable to walk up a flight of stairs without getting breathless, please do not apply for participation in this study". This will also be confirmed in the initial consultation, during which Dr. Ampat will once again ask participants this question.
* Lack of mental ability to participate in the exercise programme.
* Have had a lower-limb joint (hip or knee) replacement, as some of the exercises may be contra-indicative to these conditions.
* Participants who do not have the adequate skill of the English language - Due to lack of adequate resources and to avoid ethical issues, we will also not be including participants who do not have adequate communication skills in the English language.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Oswestry Low Back Pain Disability Questionnaire (OLBPDQ) | Baseline, 12 weeks and 6 months
  Differences in Oswestry Low Back Pain Disability Questionnaire (OLBPDQ) scores to will be assessed to quantify changes in back pain. The OLBPDQ comprises ten questions to assess the severity of back pain, and its effects on personal care, carrying out activities (walking, lifting etc.), sleep quality, social life, travelling and sex-life. Levels of pain/effects of pain will be reported by selecting one statement from five, with the most positive statement denoting a score of 0 and the most negative statement denoting a score of 5.

SECONDARY OUTCOMES:
Numerical Pain Rating Scale (NRPS) | Baseline, 12 weeks and 6 months
  Differences in 11-point Numerical Pain Rating Scale (NPRS) scores to determine changes in back pain. Participants will be required to rate their back pain on this scale, where 0 denotes 'no pain at all' and 10 denotes the 'worst possible pain'.
EuroQol 5-Dimension (EQ-5D) | Baseline, 12 weeks and 6 months
  Differences in EuroQol 5-Dimension (EQ-5D) Questionnaire scores to observe alterations in health-related quality of life
Usefulness scale for patient educational material (USE) | 12 weeks and 6 months
  Usefulness scale for patient educational material (USE) to evaluate the usefulness of the reading material provided ("Free From Pain Exercise Book" / "The Back Book"). A maximum total score of 90 suggests that the participant 'completely agrees' with nine positive statements regarding the usefullness of the information material provided, whilst a minimum score of 0 suggests that they 'completely disagree' with said statements.
Qualatitive questions | 12 weeks and 6 months
  Qualitative questions to assess participant opinions regarding the "Free From Pain Exercise Book" and "The Back Book". Questions will include 'What did you like about the "Free From Pain Exercise Book" / "The Back Book?"' and 'How do you think the "Free From Pain Exercise Book" / "The Back Book" could be improved?'.

OTHER OUTCOMES:
Compliance to participate in the "Free From Pain" exercises | 12 weeks and 6 months
  Participants in Group 1 will be required to fill in the exercise diary found at the back of the "Free From Pain Exercise Book" each time they engage in the "Free From Pain" exercises during the initial 12-week intervention period. To assess long-term compliance, they will be required to populate this second diary every time they engage in the "Free From Pain" exercises during the follow-up period.
Engagement in exercises following use of "The Back Book" | 12 weeks and 6 months
  During a phone call at 12 weeks and six months, participants in Group 2 will be asked to report how much they exercised (if at all) during the intervention and follow-up periods respectively, and what this physical activity involved.

CONTACTS AND LOCATIONS:
Overall Officials: George Ampat, MBBS, MS, FRCS, Principal Investigator — Talita Cumi Ltd.
Locations (1):
- Talita Cumi LTD., Southport, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, data will be fully anonymised. Only non-identifiable, anonymised data will be archived along with the publication for use of other researchers. For instance, the age, sex, and study results of participants will be archived indefinitely as a supplementary document to the publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available at the completion of the study on 31/12/2022. It will be available for other researchers indefinitely.
Access Criteria: The non-identifiable data will be openly available as a supplementary document to the publication.

REFERENCES:
- [Result] World Health Organisation (WHO) (2021). Musculoskeletal Conditions [Fact Sheet]. [Cited January 2021]. Retrieved from: https://www.who.int/news-room/fact-sheets/detail/musculoskeletal-conditions
- [Result] Arthritis Research UK. Understanding Arthritis: A Parliamentary Guide to Musculoskeletal Health. Chesterfield: Arthritis Research UK; 2013.
- [Result] Walker BF. The prevalence of low back pain: a systematic review of the literature from 1966 to 1998. J Spinal Disord. 2000 Jun;13(3):205-17. doi: 10.1097/00002517-200006000-00003. PMID 10872758
- [Result] Kovacs FM, Abraira V, Zamora J, Fernandez C; Spanish Back Pain Research Network. The transition from acute to subacute and chronic low back pain: a study based on determinants of quality of life and prediction of chronic disability. Spine (Phila Pa 1976). 2005 Aug 1;30(15):1786-92. doi: 10.1097/01.brs.0000172159.47152.dc. PMID 16094282
- [Result] Haas M, Groupp E, Muench J, Kraemer D, Brummel-Smith K, Sharma R, Ganger B, Attwood M, Fairweather A. Chronic disease self-management program for low back pain in the elderly. J Manipulative Physiol Ther. 2005 May;28(4):228-37. doi: 10.1016/j.jmpt.2005.03.010. PMID 15883575
- [Result] Kovacs F, Abraira V, Santos S, Diaz E, Gestoso M, Muriel A, Gil del Real MT, Mufraggi N, Noguera J, Zamora J; Spanish Back Pain Research Network. A comparison of two short education programs for improving low back pain-related disability in the elderly: a cluster randomized controlled trial. Spine (Phila Pa 1976). 2007 May 1;32(10):1053-9. doi: 10.1097/01.brs.0000261556.84266.0f. PMID 17471084
- [Result] Baker MK, Atlantis E, Fiatarone Singh MA. Multi-modal exercise programs for older adults. Age Ageing. 2007 Jul;36(4):375-81. doi: 10.1093/ageing/afm054. Epub 2007 May 30. PMID 17537741
- [Result] Campbell AJ, Robertson MC, Gardner MM, Norton RN, Tilyard MW, Buchner DM. Randomised controlled trial of a general practice programme of home based exercise to prevent falls in elderly women. BMJ. 1997 Oct 25;315(7115):1065-9. doi: 10.1136/bmj.315.7115.1065. PMID 9366737
- [Result] Cederbom S, Arkkukangas M. Impact of the fall prevention Otago Exercise Programme on pain among community-dwelling older adults: a short- and long-term follow-up study. Clin Interv Aging. 2019 Apr 26;14:721-726. doi: 10.2147/CIA.S200188. eCollection 2019. PMID 31118594
- [Result] Bystrom MG, Rasmussen-Barr E, Grooten WJ. Motor control exercises reduces pain and disability in chronic and recurrent low back pain: a meta-analysis. Spine (Phila Pa 1976). 2013 Mar 15;38(6):E350-8. doi: 10.1097/BRS.0b013e31828435fb. PMID 23492976
- [Result] Gross A, Kay TM, Paquin JP, Blanchette S, Lalonde P, Christie T, Dupont G, Graham N, Burnie SJ, Gelley G, Goldsmith CH, Forget M, Hoving JL, Bronfort G, Santaguida PL; Cervical Overview Group. Exercises for mechanical neck disorders. Cochrane Database Syst Rev. 2015 Jan 28;1(1):CD004250. doi: 10.1002/14651858.CD004250.pub5. PMID 25629215
- [Result] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Result] Young IA PT, DSc, Dunning J PT, DPT, Butts R PT, PhD, Mourad F PT, DPT, Cleland JA PT, PhD. Reliability, construct validity, and responsiveness of the neck disability index and numeric pain rating scale in patients with mechanical neck pain without upper extremity symptoms. Physiother Theory Pract. 2019 Dec;35(12):1328-1335. doi: 10.1080/09593985.2018.1471763. Epub 2018 Jun 1. PMID 29856244
- [Result] Obradovic M, Lal A, Liedgens H. Validity and responsiveness of EuroQol-5 dimension (EQ-5D) versus Short Form-6 dimension (SF-6D) questionnaire in chronic pain. Health Qual Life Outcomes. 2013 Jul 1;11:110. doi: 10.1186/1477-7525-11-110. PMID 23815777
- [Result] Holzel LP, Ries Z, Dirmaier J, Zill JM, Kriston L, Klesse C, Harter M, Bermejo I. Usefulness scale for patient information material (USE) - development and psychometric properties. BMC Med Inform Decis Mak. 2015 Apr 19;15:34. doi: 10.1186/s12911-015-0153-7. PMID 25927192